CLINICAL TRIAL: NCT02889848
Title: An Open Label, Dose Escalation Study to Assess Safety and Tolerability of Collagenase Clostridium Histolyticum (EN3835) in Subjects With Uterine Leiomyoma (Fibroids)
Brief Title: Safety and Tolerability of Collagenase Clostridium Histolyticum (EN3835) to Treat Uterine Leiomyoma (Fibroids)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Advance Biofactures Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIB1154
Record Dates: First submitted 2016-08-22; First posted 2016-09-07 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2018-06

CONDITIONS: Fibroids, Uterine; Leiomyoma
MeSH Terms: conditions — Leiomyoma | interventions — Sodium Chloride; Microbial Collagenase

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (5):
- Saline only (Sham Comparator): Injection of saline to assess the injection procedure
  Interventions: Other: Saline
- 1.16 mg EN3835 (Experimental): Injection of maximum marketed dose of EN3835 regardless of fibroid size
  Interventions: Drug: EN3835
- Dose 1 (Experimental): Injection of 0.05 mg EN3835 per cm3 fibroid
  Interventions: Drug: EN3835
- Dose 2 (Experimental): Injection of 0.1 mg EN3835 per cm3 fibroid
  Interventions: Drug: EN3835
- Dose 3 (Experimental): Injection of 0.2 mg EN3835 per cm3 fibroid
  Interventions: Drug: EN3835

INTERVENTIONS:
Other: Saline — Saline injection
  Arms: Saline only
Drug: EN3835 — Comparison of maximum marketed dose and multiple doses EN3835
  Other Names: Collagenase clostridium histolyticum
  Arms: 1.16 mg EN3835; Dose 1; Dose 2; Dose 3

SUMMARY:
This pilot study evaluates the safety and tolerability of a single injection of collagenase enzyme directly into a uterine fibroid in subjects already selected for hysterectomy or myomectomy.

Fibroids contain excessive amounts of collagen and it is possible that digestion of collagen may be beneficial in reducing pain and bleeding associated with fibroids.

Three subjects will be injected with saline only to evaluate the safety and effectiveness of the injection method. Additional subjects will then be injected with increasing doses of study drug.

DETAILED DESCRIPTION:
Collagenase enzyme breaks down collagen and has shown efficacy in clinical trials for a number of diseases for which there is an accumulation of collagen.

It is possible that lysis of collagen may reduce the collagen content of fibroids thus decreasing the size of fibroids, and possibly reducing the stiffness of fibroids. This may result in reducing the symptoms of pain and bleeding associated with fibroids.

In this study three subjects will be injected with saline only followed immediately by hysterectomy in order to evaluate the safety and effectiveness of the injection method.

Twelve subjects will receive a single injection of study drug as follows: three subjects will receive a set dose of collagenase enzyme followed by hysterectomy or myomectomy 24-96 hours later (Group 1) to evaluate safety of the injection of study drug. Nine subjects will then receive increasing doses of collagenase enzyme followed by hysterectomy or myomectomy 60-90 days later (Group 2).

ELIGIBILITY:
Inclusion Criteria:

* Parous and non-parous women who have completed child-bearing (age criteria of > 35 years-old, and <50 years-old)
* Currently practicing or willing to practice contraception throughout the duration of the study
* Women with at least one or two fibroids greater than or equal to 3 cm diameter, and less than or equal to 10 cm diameter for subjects in Group 1, and at least one fibroid greater than or equal to 3 cm diameter, and less than or equal to 10 cm diameter for subjects in Group 2
* Fibroids will be intramural fibroids which will be surrounded by a layer of myometrium. Fibroids must be well visualized on ultrasound examination and provide a clear path for injection
* Women who were planning to undergo abdominal hysterectomy or myomectomy for treatment of symptomatic fibroids. Subjects must be willing to defer the operation until 24-96 hours after study treatment for Group 1 and for 60-90 days after study treatment for Group 2. The patients will understand that they may choose to have surgery or any other non-study treatment at any time after enrollment and end study participation
* "Typical" large fibroids visualized as hypo-intense on a T2-weighted MRI scan

Exclusion Criteria:

* Inability to understand study procedures or to comply with study visits and requirements
* BMI > 40kg/m2
* History of allergic reaction to study medication (Collagenase Clostridium Histolyticum) or any components of the study drug
* Inability to undergo hysterectomy or myomectomy
* Inability to tolerate MRI and transvaginal ultrasound procedures (i.e. presence of an intra-uterine device (IUD), pacemakers, aneurismal clips or other metallic devices that are not compatible with magnetic resonance imaging). However women with IUD's compatible with MRI are eligible for the study
* Medical problems including: genetic diseases that cause fibroids, history of thromboembolic (blood clot) events or need for anticoagulation (Coumadin, Heparin, etc.) Subjects taking or planning to take anti-coagulant medication (except for ≤ 150 mg aspirin daily) within 7 days administration study drug and within 7 days before and after hysterectomy
* A history of cancer within the past 5 years
* Abnormal liver function tests (typically, will be >20% elevation). Mild elevations will be at the discretion of the investigators, but undiagnosed liver conditions will represent an exclusion criterion
* Pregnancy or lactation. Pregnancy will be evaluated by urine test every 30 days if necessary. Patients will be asked to use non-hormonal contraception methods while in this study
* Severe anemia (hematocrit <30). Mild anemia is common in women with fibroids
* Recent rapid growth of fibroids (i.e. doubling in size within one-six months period)
* Any use of agents like Imidazoles, due to possible interference with metabolism
* Unevaluated gynecologic abnormalities (unexplained vaginal bleeding, cervical dysplasia, or abnormal adnexal/ovarian mass)
* Fibroids that are visualized on T2 and T1 weighted MRI as hyperdense or show cystic degeneration
* Inability to undergo injection of fibroid with study drug for any reason, anatomic or other
* Has a known systemic allergy to collagenase or any other excipient of EN3835 or any other procedural medication
* Has, at any time, received collagenase as a treatment
* Is planning to be treated with commercial XIAFLEX at any time during the study
* Type 0 submucosal fibroids, submucosal fibroids with significant protrusion/ pedunculation and subserosal fibroids are not appropriate candidates for the injections

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events following a single injection of EN3835 into a fibroid | Through hysterectomy or myomectomy (average = 60-90 days post injection)
  Assessed by number of subjects with uterine injury or peritoneal irritation determined post hysterectomy

SECONDARY OUTCOMES:
Change in symptoms of pain and bleeding and quality of life | Throughout the study prior to hysterectomy or myomectomy(avg 60-90 days post injection study drug)
  Determined by standardized questionnaires for menstrual distress, quality of life and sexual activity; McGill Pain Questionnaire
Reduction in size of treated fibroids- Group 2 | 60-90 days post injection study drug
  Size of fibroid to be determined post hysterectomy or myomectomy
Increased rate of apoptosis of treated fibroids -Group 2 | 60-90 days post injection study drug
  Specimens to be taken post hysterectomy or myomectomy and evaluated by TUNEL staining
Reduction in collagen content of treated fibroids-Group 2 | 60-90 days post injection study drug
  Specimens to be taken post hysterectomy or myomectomy and by tested histology stains
Reduction in stiffness of treated fibroid-Group 2 | 60-90 days post injection study drug
  Specimens to be taken post hysterectomy or myomectomy and tested via rheometry

CONTACTS AND LOCATIONS:
Overall Officials: James Segars, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Islam MS, Afrin S, Singh B, Jayes FL, Brennan JT, Borahay MA, Leppert PC, Segars JH. Extracellular matrix and Hippo signaling as therapeutic targets of antifibrotic compounds for uterine fibroids. Clin Transl Med. 2021 Jul;11(7):e475. doi: 10.1002/ctm2.475. PMID 34323413